CLINICAL TRIAL: NCT06378645
Title: Prospective, Randomized-Controlled Study of the Effect of Propofol vs. Sevoflurane on Erections During Narcosis in Transurethral Surgery
Brief Title: Effect of Propofol vs. Sevoflurane on Erections During Narcosis In Transurethral Surgery
Acronym: PENIS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Etienne Xavier Keller (Other)
Responsible Party: Sponsor-Investigator, Etienne Xavier Keller, Assistant Professor, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023-01682
Record Dates: First submitted 2024-04-15; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Erection; Incomplete
Keywords: transurethral surgery; penile tumescence; intraoperative erection; propofol; sevoflurane; investigator initiated trial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The authorized study nurse will hand the upcoming envelope with the treatment allocation to the anesthesiologist. The patient and the urologists (who is measuring the outcome) will not know which form of general anesthesia will be performed. Herewith, blankets in the operating room will hide installations used by the anesthesiologists to prevent the urologists witnessing the assigned narcosis form. Before the surgical sign-out, while still scrubbed in and with the patient under anesthesia, the anesthesiologists will ask the urologists about the outcome questionnaire. Together, they will fill in the paper case report form (CRF).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group: Propofol (Active Comparator): The patients in the intervention group are receiving a general anesthesia with Propofol.
  Interventions: Drug: General Anesthesia: Propofol
- Control group: Sevoflurane (Active Comparator): The patients in the control group are receiving a general anesthesia with Sevoflurane.
  Interventions: Drug: General Anesthesia: Sevoflurane

INTERVENTIONS:
Drug: General Anesthesia: Propofol — Transurethral surgery at the Department of Urology (University Hospital Zurich) performed under study arm-specific anesthesia.
  Propofol will be administered intravenously using the target-controlled infusion algorithm with effect site concentrations between 1.5-4.0 µg/ml necessary.
  Arms: Intervention group: Propofol
Drug: General Anesthesia: Sevoflurane — Transurethral surgery at the Department of Urology (University Hospital Zurich) performed under study arm-specific anesthesia.
  Sevoflurane will be given in gaseous form via the endotracheal tube in concentrations between 1.5-2.5% Vol.
  Arms: Control group: Sevoflurane

SUMMARY:
Penile erection is an unwanted event in transurethral (through the urethra) surgeries, which may be associated with adverse outcomes such as impaired access, prolonged operation time, the need to abort the operation, or the necessity for ancillary measures to achieve penile flaccidity, such as the injection of certain medications directly into the penis.

To reduce greenhouse gas emissions, the primary use of propofol instead of gaseous agents is being recommended for general anesthesia. Whether propofol may be associated with an increased or decreased rate of unwanted intraoperative penile erection compared to other anesthetic agents is not known. More generally, there are no high-quality studies available to evaluate the impact of the type of general anesthesia on the risk of unwanted penile erections during surgery.

This study aims to determine whether general anesthesia with propofol is more likely to cause intraoperative erections compared to sevoflurane during transurethral operations.

DETAILED DESCRIPTION:
Introduction

Intraoperative penile erection is an unwanted event during transurethral surgery, since it may impair the access to the urinary pathways thus prolonging operation time and sometimes requiring ancillary measures to reach penis flaccidity. Ultimately, penile erections may cause operation abortion. Fortunately, reversal of penile erections can be achieved intraoperatively by pharmacological interventions such as intravenous administration of ketamine or intracorporeal injection of vasoactive agents such as phenylephrine or epinephrine, although these medications are in turn associated with potentially severe secondary effects. The incidence of intraoperative penile erections is reported to lay between 2.2% and 3.5% in adults. The evidence on the topic is of limited quality, thus the risk factors and frequency of unwanted penile erections in transurethral interventions remain to be evaluated.

The use of propofol has been associated with a particularly high risk for sexual arousal and intraoperative erections, reaching an incidence of unwanted erections of up to 10% in pediatric case series undergoing urethral surgery. The causes and the pathophysiology have been partially explored, although the leading mechanisms remain debated.

In an effort to reduce greenhouse gas emissions, the primary use of propofol instead of gaseous agents for general anesthesia has been introduced at our tertiary academic hospital in October 2022. This institutional change in anesthesia protocol has led to a perceived increase in the rates of unwanted intraoperative erections and interventions to achieve penile flaccidity, possibly associated with the increased use of propofol. Because there are no high-quality studies investigating the impact of various anesthetic agents on penile tumescence in men during transurethral procedures in literature to date, anesthesiologist and urologist at our institution initiated together a prospective randomized controlled trial comparing the incidence of intraoperative penile tumescence during propofol versus sevoflurane general anesthesia.

Sample size determination

The investigators anticipate the detection of a 9% points absolute risk elevation of intraoperative erections in the intervention group (propofol) compared to the control group (sevoflurane). To detect a 9% risk elevation, which is considered a clinically relevant increase in the intervention group (10% anticipated) in comparison with the control group (1% anticipated), and to assure a study power of 80% with dichotomous outcome variable and a 2-sided significance level of alpha = 0.05, 100 patients will be needed in each group (200 patients in total). The calculated sample size is appropriate to the hypothesis being tested, so that any results will be appropriately generalizable.

Statistical methods

Prior to data export, a statistical analysis plan will be written up and signed by the principle investigator and the trial statistician. The analysis will be performed blinded and using dynamic reporting tools in a fully scripted way to guarantee highest standards regarding reproducibility. The primary analysis of the primary outcome will be performed using a logistic regression model with logit link function with treatment group, as well as the stratification variable as an independent variable. The effect measure will be an odds ratio.

Enrolment and study schedule

Every male patient referred for surgical consultation prior to transurethral surgery will be screened by age and International Index of Erectile Function:5-item version (IIEF-5) score. If the patient is eligible for participation in the study, he will be informed accordingly. After giving his informed consent, patients will be randomized to the intervention or control group by computerized random sequence generation on the day of surgery. Within one day after the intervention, patients will be visited by the urology and anesthesiology team at the end of study.

Data collection

The following parameters will be recorded for each patient: age, blood pressure, heart rate, weight, height, IIEF-5 Score as well as the duration of, reason for and the type of transurethral intervention. All primary and secondary outcomes will be reported immediately prior to the operation's sign-out by the operating urologists. Until the end of the study visit, all patients will be screened for related adverse events (AEs). In the case of an AE, the type of AE, grade of AE, and time until resolution of AE will be recorded. All parameters are entered into a secure electronic database.

Auditing, Data monitoring and Harms

Regular monitoring visits will be performed prior to the start and during the period of the study at the investigator's site. During internal audits, all paper CRF and the electronical database will be inspected. Since both anesthesiological drugs are licensed for their use, a continues data monitoring board will be not be necessary and no interim analysis is planned, in accordance with local laws and ethical principles. Any complication of the investigational drugs will be collected as a secondary outcome, as detailed above.

Consent

All patients will be informed about the study by trained urologists and anesthesiologists. Patient inclusion into the study will only occur after written consent of the patient has been obtained. When the participant withdraws consent, data collected prior to the date of withdrawal remains within the electronical study database and can be included in data analysis. Participants who discontinue the study prior to data collection will be replaced. Individual medical information obtained within this study is considered confidential and disclosure to third parties is prohibited. Subject confidentiality will be further ensured by utilizing patient identification code to correspond to treatment data in the computer files. For source data verification purposes, authorized representatives of the investigator, a competent authority or monitoring may require direct access to parts of the medical records relevant to the study, including participants' medical history. The planned clinical trial entails only minimal risks for study participants considering that both investigated drugs are licensed for use by the Swiss medical authorities and have been regularly used in daily routine for many years.

ELIGIBILITY:
Inclusion Criteria:

* Planned transurethral operation in the department of urology.
* Preoperative IIEF-5 Score ≥12
* Planned surgery time ≥15min

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Inability to provide informed consent.
* Contraindications to Propofol or Sevoflurane, e.g. known hypersensitivity or allergy.
* Known or suspected non-compliance, drug or alcohol abuse.
* Participation in another study with an investigational drug within the 30 days preceding and during the present study.
* Previous enrolment into the current study.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Penile Erection | Assessment during the operation and reporting before the end of the surgery.
  The primary endpoint "penile erection" will be analyzed as a binary outcome flaccid or erect. The occurrence of an erect penis at any time during surgery is classified as erect penile tumescence. Flaccid penile tumescence is classified only if erect penile tumescence does not occur at any point during the operation. The beginning and end of the operation are defined as the first insertion and last retrieval of all instruments, respectively. The penile tumescence will be reported in a simplified version of the validated EHS (erection hardness score): 0: flaccid, 1: increased tumescence, but not fully erect, 2: full erection.
  Erect penile tumescence is defined as achieving a score of either 1 or 2, whereas flaccid penile tumescence is defined as a score of 0.

SECONDARY OUTCOMES:
Prolongation of the surgery | Assessment during the operation and reporting before the end of the surgery.
  The treating urologist will answer a questionnaire specifying if there was a subjective prolongation of the surgery (yes (time)/no).
Change in operative strategy | Assessment during the operation and reporting before the end of the surgery.
  The treating urologist will answer a questionnaire specifying if there was a change in operative strategies due to penile tumescence (yes/no).
Adaptions of instruments or approaches | Assessment during the operation and reporting before the end of the surgery.
  The treating urologist will answer a questionnaire immediately after the surgery specifying if there were adaptions of instruments or approaches due to penile tumescence (yes/no).
Altered operative outcome | Assessment during the operation and reporting before the end of the surgery.
  The treating urologist will answer a questionnaire specifying if there was a change of the operative outcome due to penile tumescence (yes/no).
Necessity for a drug application to decrease penile tumescence | Assessment during the operation and reporting before the end of the surgery.
  The treating urologist will answer a questionnaire specifying if there was a necessity for a drug application to decrease penile tumescence? (Yes: 1. ketamine bolus; 2. Intracorporal Injection of phenylephrine, No)
Complications arisen | Assessment for 24 hours after the surgery.
  The treating urologist will answer a questionnaire specifying if there were complications due to an intraoperative erection of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne X Keller, Ass Prof, MD, Principal Investigator — University Hospital Zurich, University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
After successful publishing, the data will be made available in anonymized form stored and in an open-access repository.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: After successful publishing
Access Criteria: After successful publishing

REFERENCES:
- [Derived] Scherer TP, von Deschwanden C, Held U, Poyet C, Kwok JL, Kandler L, Schlapfer M, Keller EX, Schmid FA. Effect of Propofol Versus Sevoflurane on Erections during Narcosis in Transurethral Surgery: The PENIS Trial. Eur Urol Open Sci. 2024 Sep 24;69:100-104. doi: 10.1016/j.euros.2024.08.021. eCollection 2024 Nov. PMID 39381594